CLINICAL TRIAL: NCT05811234
Title: An International, Prospective, Observational Cohort Study to Assess Patient Treatment Satisfaction, Patient-reported Outcomes, Effectiveness, and Safety of a Fixed-dose Combination of Calcipotriene/Betamethasone Dipropionate PAD Cream in the Treatment of Mild-to-moderate Plaque Psoriasis of the Scalp in Adults (PRO-SCALP)
Brief Title: A Study to Assess Treatment Satisfaction, Patient-reported Outcomes, Effectiveness, and Safety of a Fixed-dose Combination of Calcipotriene/Betamethasone Dipropionate PAD Cream in the Treatment of Mild-to-moderate Plaque Psoriasis of the Scalp in Adults
Acronym: PRO-SCALP
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M-22201-41
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis
Keywords: Mild-to-moderate plaque psoriasis; Prospective; Psoriasis; PRO-SCALP; Plaque psoriasis of the scalp
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAL/BDP PAD Cream:: Participants who have been prescribed CAL/BDP PAD cream treatment to manage plaque psoriasis of the scalp according to summary of product characteristic (SmPC) in routine clinical practice settings will be observed prospectively for up to 8-12 weeks.
  Interventions: Drug: CAL/BDP PAD Cream

INTERVENTIONS:
Drug: CAL/BDP PAD Cream — As provided in real-world clinical practice.
  Other Names: Wynzora®

SUMMARY:
The main aim of this study is to assess treatment satisfaction, quality of life, treatment preference, adherence and convenience, psychosocial effects of scalp psoriasis, sleep quality, and effectiveness, and safety of Calcipotriene/Betamethasone Dipropionate (CAL/BDP) PAD cream in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (greater than or equal to [>=] 18 years) male or female participants with mild-to-moderate plaque psoriasis of the scalp (defined as scalp-PGA score of 2 or 3 at baseline) with or without involvement of the trunk and limbs, and who may or may not have been previously treated (treatment-naive participants) with other anti-psoriatic therapies.
2. Participants who have been prescribed CAL/BDP PAD cream (Wynzora®) treatment to manage plaque psoriasis of the scalp according to SmPC in routine clinical practice.
3. Willingness and ability to participate in the study; participants must give their written consent to participate.

Exclusion Criteria:

1. Participants with severe plaque psoriasis, per physician global assessment.
2. Participants with erythrodermic, exfoliative or pustular psoriasis.
3. Participants previously treated with systemic drugs for psoriasis (conventional or biologic) within the last 12 weeks prior to inclusion.
4. Concomitant systemic treatment with anti-psoriatic drugs.
5. Concomitant treatment of any type for plaque psoriasis of the scalp.
6. Hypersensitivity to the active substances or to any of the excipients of CAL/BDP PAD cream (Wynzora®).
7. Participants with known disorders of calcium metabolism.
8. Participants with viral (e.g., herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, skin manifestations in relation to tuberculosis, perioral dermatitis, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne vulgaris, acne rosacea, rosacea, ulcers, and wounds.
9. Pregnant or breastfeeding women, except when the potential benefit justifies the potential risk.
10. Participants unable to comply with the requirements of the study or who in the opinion of the study physician should not participate in the study.
11. Participants for whom medical chart is inaccessible to physicians to complete baseline data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female participants with mild-to-moderate plaque psoriasis of the scalp will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- Germany (11):
  - DE12, Ahaus
  - DE07, Augsburg
  - DE06, Cologne
  - DE08, Freising
  - DE10, Mainz
  - DE01, Mannheim
  - DE05, Mölln
  - DE03, Mönchengladbach
  - DE04, Pforzheim
  - DE02, Potsdam
  - DE11, Remscheid
- Spain (13):
  - ES04, Alcorcón
  - ES10, Badalona
  - ES02, Barcelona
  - ES06, Barcelona
  - ES09, Barcelona
  - ES05, Bilbao
  - ES03, Granollers
  - ES07, Lleida
  - ES08, Pontevedra
  - ES12, Salamanca
  - ES11, Seville
  - ES13, Seville
  - ES01, Zaragoza
- United Kingdom (13):
  - UK10, Blackburn
  - UK02, Chertsey
  - UK06, Chipping Norton
  - UK08, Cockermouth
  - UK03, Crewe
  - UK07, Exeter
  - UK14, Glasgow
  - UK15, Kirkcaldy
  - UK11, Leicester
  - UK01, London
  - UK05, Saint Neots
  - UK04, Salisbury
  - UK12, Wellingborough

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 sites across three European countries (Germany, Spain, and the United Kingdom) from 13 June 2023 to 01 October 2024.
Pre-assignment Details: A total of 291 participants were enrolled in this study.
Groups:
- CAL/BDP PAD Cream: Participants who have been prescribed a fixed dose of Calcipotriene/Betamethasone Dipropionate PAD cream (CAL/BDP PAD cream) treatment to manage plaque psoriasis of the scalp according to summary of product characteristic (SmPC) in routine clinical practice settings were observed for up to 8-12 weeks.
Period: Overall Study
Arm/Group | CAL/BDP PAD Cream
Started | 291
Safety Population (Safety population included all participants for whom it is known that they had at least one CAL/BDP PAD cream application during the study observation period.) | 291
Full Analysis Set (FAS) (FAS included all those participants in the safety population that had at least one post-baseline assessment* for primary endpoint.) | 253
Completed | 265
Not Completed | 26
Not completed — Loss of Effectiveness | 2
Not completed — Adverse Event | 4
Not completed — Pregnancy | 1
Not completed — Disease progression | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 13
Not completed — Personal reason, or the patient stops taking the study treatment | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants for whom it is known that they had at least one CAL/BDP PAD cream application during the study observation period.
Arm/Group | CAL/BDP PAD Cream
Number analyzed (Participants) | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.88 (17.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity were not collected from any participant.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 265
  More than one race | 8
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Absolute Treatment Satisfaction Questionnaire for Medication Version 9 (TSQM-9) Domain Total Score at Week 12
Description: TSQM-9 was a 9-item clinically validated psychometric instrument developed from the TSQM 1.4. TSQM-9 measures participant satisfaction with the medication in 3 domains: Effectiveness, convenience, and global satisfaction. The scores were computed by adding items for each domain, i.e., 1 to 3 for effectiveness, 4 to 6 for convenience, and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) x 3 items = 18 for effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100, with higher scores indicating greater satisfaction for that domain.
Time Frame: At end of study observation period (Week 12)
Population: FAS included all those participants in the safety population that had at least one post-baseline assessment for primary endpoint.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CAL/BDP PAD Cream
Number analyzed (Participants) | 253
Score on a scale
  Effectiveness Total Score: At Week 12 | 73.56 [70.41 to 76.71]
  Convenience Total Score: At Week 12 | 72.07 [69.65 to 74.49]
  Global Satisfaction Total Score: At Week 12 | 75.97 [73.30 to 78.65]

2. Secondary Outcome: Absolute Scalpdex Questionnaire Domine (Symptoms, Emotions, and Functioning) Scores
Description: Scalpdex is a scalp dermatitis-specific quality of life (QoL) instrument that can be used to determine which aspect of the disease most bothers the participant and to evaluate QoL as one variable of responsiveness to the therapeutic intervention. It has 23 items, with possible answers scoring on a 5-point Likert-type scale of 0 to 100 ("never" = 0, "rarely" = 25, "sometimes" = 50, "often" = 75, and "all the time" = 100). The final domine scores (symptoms, emotions, and functioning) are calculated by the mean of the item scores pertaining to each scale is the average of the scores of the 23 items with range of 0 to 100. A lower score on symptoms, emotions, and functioning represents a better related-QoL for each scale.
Time Frame: At end of study observation period (Week 12)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CAL/BDP PAD Cream
Number analyzed (Participants) | 253
Score on a scale
  Symptoms: At Week 12 | 22.66 [20.37 to 24.95]
  Emotions: At Week 12 | 29.53 [27.08 to 31.99]
  Functioning: At Week 12 | 26.88 [24.22 to 29.53]

3. Secondary Outcome: Percentage of Participants Achieved Scalp Physician's Global Assessment (Scalp-PGA) Treatment Success at Week 4 and 12
Description: Scalp-PGA treatment success was defined as a scalp-PGA score of 0 (clear) or 1 (almost clear) and with a minimum 2 points improvement from baseline, on the scalp.
Time Frame: At Week 4 and End of study observation period (Week 12)
Population: FAS included all those participants in the safety population that had at least one post-baseline assessment for primary endpoint. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies who were evaluable at specific timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | CAL/BDP PAD Cream
Number analyzed (Participants) | 250
Percentage of participants
  Scalp-PGA Success at Week 4: Yes: number analyzed (Participants) | 25
  Scalp-PGA Success at Week 4: Yes | 48.00
  Scalp-PGA Success at Week 4: No: number analyzed (Participants) | 25
  Scalp-PGA Success at Week 4: No | 52.00
  Scalp-PGA Success at Week 12: Yes | 68.40
  Scalp-PGA Success at Week 12: No | 31.60

4. Secondary Outcome: Absolute Scalp Worst Itch Numerical Rating Scale (WI-NRS) Questionnaire Score
Description: WI-NRS is a self-administered scale to assess participants worst level of itching on the scalp (in the last week). The scale has a single-item that describes the worst level of itching on the scalp due to psoriasis in the last week on an 11-point scale anchored at 0 (no itching) and 10 (worst itching imaginable).
Time Frame: Baseline, End of study observation period (Week 12)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CAL/BDP PAD Cream
Number analyzed (Participants) | 253
Score on a scale
  Baseline | 6.43 [6.13 to 6.73]
  At Week 12 | 2.66 [2.34 to 2.97]

ADVERSE EVENTS:
Time Frame: Baseline up to end of study observation period (Week 12)
Arm/Group | CAL/BDP PAD Cream
All-Cause Mortality (participants affected / at risk) | 1/291
Serious Adverse Events (participants affected / at risk) | 2/291
Other Adverse Events (participants affected / at risk) | 13/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAL/BDP PAD Cream (N=291)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAL/BDP PAD Cream (N=291)
Conjunctivitis (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 2
Urticaria Chronic (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT05811234/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT05811234/SAP_001.pdf